CLINICAL TRIAL: NCT00596089
Title: Use of Jumping Mechanography as a Method to Assess Musculoskeletal Status in Older Adults: A Pilot Study
Brief Title: Use of Jumping Mechanography as a Method to Assess Musculoskeletal Status in Older Adults
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-0274
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2008-01

CONDITIONS: Musculoskeletal Status; Muscle Weakness
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Men and women 60 years and older
- 2: Men and women 20-30 years of age

SUMMARY:
Decline in muscle function may increase risk of hip fracture and decrease quality of life. Different tests are currently used to measure muscle function but they do not work for all individuals. A test called "jumping mechanography," which measures jumping power, may be useful in more people and obtain better information. This study will help us determine whether this test is able to detect differences between muscle function in younger and older adults, as well as whether it is a safe method to use in all ages.

ELIGIBILITY:
Inclusion Criteria:

1. Women and men aged 20 to 30 or ≥ 60 years
2. Able and willing to sign informed consent.
3. Ability to stand without assistance.

Exclusion Criteria:

1. Acute pain different and/or worse than the individuals chronic baseline pain
2. History of recent trauma to musculoskeletal system
3. Neuromuscular disease impairing balance to the degree of not being able to stand without assistance.
4. History of fragility fracture within the last year
5. Patients with a BMD T-score of less than -3.5 at any measured site and a vertebral fracture.
6. History of severe end-organ disease, e.g., cardiovascular, hepatic, hematologic, pulmonary, etc., which might limit the ability to complete this study.
7. Recent history of malignancy with metastasis to the musculoskeletal system.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women 60 years and older and men and women 20-30 years of age
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the instantaneous weight corrected peak power taken from the maximal countermovement jump | single session

CONTACTS AND LOCATIONS:
Overall Officials: Neil C Binkley, MD, Principal Investigator — University of Wisconsin - Institute on Aging
Locations (1):
- University of Wisconsin Osteoporosis Clinical and Research Program, Madison, Wisconsin, United States